CLINICAL TRIAL: NCT04160546
Title: Multicenter, Open-Label, Single Arm, Phase II Exploratory Study to Evaluate the Reinduction and Second Stop of TKI with Ponatinib in CML in Molecular Response (ResToP)
Brief Title: Study to Evaluate the Reinduction and Second Stop of TKI with Ponatinib in CML in Molecular Response (ResToP)
Acronym: ResToP
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion CRIS de Investigación para Vencer el Cáncer (Other)
Collaborators: Incyte Biosciences UK (Industry); Apices Soluciones S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ResToP; 2018-003281-14 (EudraCT Number); 2023-508993-27-00 (EU CTIS Number)
Record Dates: First submitted 2019-11-08; First posted 2019-11-13 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Chronic Myeloid Leukemia, Chronic Phase
Keywords: Chronic Myeloid Leukemia; Ponatinib
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ponatinib plus ASA treatment (Experimental): Patients will be treated with ponatinib 15 mg/day plus 100 mg/day ASA for 104 weeks. After that, ponatinib and ASA will be stopped.
  Interventions: Drug: Ponatinib 15 MG; Drug: Acetylsalicylic acid 100 MG

INTERVENTIONS:
Drug: Ponatinib 15 MG — Patients will receive ponatinib 15 mg/day for 104 weeks orally. Ponatinib will be self-administered by the patient on a daily schedule.
  Acetyl salicylic acid (ASA) (100 mg) will be used such auxiliary medicinal product in order to prevent vascular occlusive events related with ponatinib.
Drug: Acetylsalicylic acid 100 MG — Patients will receive acetylsalicylic acid 100 mg/day for 104 weeks orally.

SUMMARY:
The purpose of the present study is to determine the rate of successful treatment-free remission (TFR) within the first 52 weeks following cessation of ponatinib treatment in patients who achieved MR4. Eligible patients had been previously treated with TKI and when patients achieved an optimal molecular response, TKI treatment was discontinued. After loss of response, patients were treated again with a TKI treatment and have documented MR4 for one year at the time of switch to ponatinib to study entry. MR4 is defined as BCR-ABL transcript level ≤ 0.01% IS or undetectable BCR-ABL levels with sample sensitivity of at least 4 log.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age.
2. ECOG Performance Status of 0, 1, or 2.
3. Patient with diagnosis of BCR-ABL positive and Ph+ CML-Chronic Phase.
4. Patients who failed the first attempt of TKI discontinuation and after TKI reintroduction they achieve again MR4 and it is maintained and confirmed for more than one year.
5. Patients who are able to take oral therapy
6. Adequate end organ function as defined by:

   1. Direct bilirubin ≤ 1.5 x ULN except for i) patient with documented Gilbert's syndrome for whom any bilirubin value is allowed and ii) for patients with asymptomatic hyperbilirubinemia (liver transaminases and alkaline phosphatase within normal range),
   2. SGOT(AST) and SGPT(ALT) ≤ 2.5 x ULN,
   3. Serum lipase and amylase ≤ 1.5 x ULN,
   4. Alkaline phosphatase ≤ 2.5 x ULN,
   5. Serum creatinine ≤ 1.5 x ULN.
7. Patients must have the following electrolyte values ≥ LLN limits or corrected to within normal limits with supplements prior to the first dose of study medication:

   1. Potassium,
   2. Magnesium,
   3. Total calcium (corrected for serum albumin)
8. Patients must have normal marrow function as defined below:

   1. Absolute Neutrophil Count (ANC) ≥ 1.5 x 109/L,
   2. Platelets ≥ 100 x 109/L.
   3. Hemoglobin > 9 g/dL.
9. Patients with preexisting, well-controlled diabetes can be included.
10. Have normal QTcF interval on screening ECG evaluation, defined as QTcF of ≤ 450 ms in males or ≤ 470 ms in females.
11. Have a negative pregnancy test documented prior to enrollment (for females of childbearing potential).
12. Be willing and able to comply with scheduled visits and study procedures.
13. Patients with the ability to comprehend and sign the informed consent.
14. Written informed consent obtained prior to any screening procedures.

Exclusion Criteria:

1. Prior accelerate phase, blast crisis or autologous or allogenic transplant.
2. Patients with known atypical transcript. An atypical transcript is defined by the presence of any transcript in the absence of the major transcripts b3a2 (e14a2) and b2a2 (e13a2) or p210 protein.
3. CML treatment resistant mutation(s) (T315I, E255K/V, Y253H, F359C/V) detected if a testing was done in the past (there is no requirement to perform mutation testing at study entry if it was not done in the past).
4. Are taking medications with a known risk of torsades de pointes (Annex 5).
5. Patient ever attempted to permanently discontinue TKI treatment.
6. Severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol (e.g., uncontrolled diabetes (defined as HbA1c > 9%), uncontrolled infection).
7. Have clinically significant, uncontrolled, or active cardiovascular disease, specifically including, but not restricted to:

   1. Any history of MI, unstable angina, cerebrovascular accident, or TIA.
   2. Any history of peripheral vascular infarction, including visceral infarction.
   3. Any revascularization procedure, including the placement of a stent.
   4. Congestive heart failure (NYHA class III or IV) within 6 months prior to enrollment, or LVEF less than lower limit of normal, per local institutional standards, within 6 months prior to enrollment.
   5. History of clinically significant (as determined by the treating physician) atrial arrhythmia or any history of ventricular arrhythmia.
   6. Venous thromboembolism, including deep venous thrombosis or pulmonary embolism, within 6 months prior to enrollment.
8. Have uncontrolled hypertension (diastolic blood pressure > 90 mmHg; systolic > 150 mmHg). Patients with hypertension should be under treatment on study entry to effect blood pressure control.
9. Have a history of alcohol abuse.
10. History of acute pancreatitis within 1 year prior to study entry or past medical history of chronic pancreatitis.
11. Have malabsorption syndrome or other gastrointestinal illness that could affect oral absorption of study drug.
12. Known presence of a significant congenital or acquired bleeding disorder unrelated to cancer.
13. Have a history of another malignancy, other than cervical cancer in situ or no metastatic basal cell or squamous cell carcinoma of the skin; the exception is if patients have been disease-free for at least 5 years, and are deemed by the investigator to be at low risk for recurrence of that malignancy.
14. Have undergone major surgery (with the exception of minor surgical procedures, such as catheter placement) within 14 days prior to first dose of ponatinib.
15. Treatment with other investigational agents (defined as not used in accordance with the approved indication) within 4 weeks of Day 1.
16. Patients actively receiving therapy with strong CYP3A4 inhibitors and/or inducers, and the treatment cannot be either discontinued or switched to a different medication prior to study entry. See Annex 6 for a list of these medications. This list may not be comprehensive.
17. Patients actively receiving therapy with herbal medicines that are strong CYP3A4 inhibitors and/or inducers, and the treatment cannot be either discontinued or switched to a different medication prior to study entry. These herbal medicines may include Echinacea (including E. purpurea, E. angustifolia and E. pallida), Piperine, Artemisinin, Hyperico, and Ginkgo.
18. Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either safely discontinued or switched to a different medication prior to study entry.
19. Have an ongoing or active infection; this includes, but is not limited to, the requirement for intravenous antibiotics.
20. Have a known history of human immunodeficiency virus infection; testing is not required in the absence of prior documentation or known history.
21. Have hypersensitivity to the ponatinib active substance or to any of its inactive ingredients.
22. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
23. Patients must not have a contraindication or a known hypersensitivity to ASA.
24. Patients with rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption.
25. Patients with previous or current hepatitis B virus infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-17 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a maintained MMR within 52 weeks following ponatinib Treatment-Free Remission (TFR) | 52 weeks
  This variable is defined as the number of patients who have a maintained MMR and have not restarted TKI therapy in the first 52 weeks after starting ponatinib TFR phase divided by the number of patients who entered ponatinib TFR phase.

SECONDARY OUTCOMES:
Evaluate the toxicity and safety profile of 15 mg/24h dose treatment of ponatinib combined with ASA. | 104 weeks
  The number and percentage of patients with treatment-emergent adverse events (new or worsening from baseline) will be summarized by system organ class (SOC) and/or preferred term (PT), severity (based on CTCAE grades), type of adverse event and relation to study treatment.
Evaluate thromboembolic events for study period. | 104 weeks
  The number and percentage of patients with thromboembolic events will be summarized by preferred term, severity (based on CTCAE grades), type of adverse event, relation to study treatment by the phases or subsets previously described.
Evaluate hemorrhagic events for study period. | 104 weeks
  The number and percentage of patients with hemorrhagic events will be summarized by preferred term, severity (based on CTCAE grades), type of adverse event, relation to study treatment by the phases or subsets previously described.
Evaluate hemolytic events for study period. | 104 weeks
  The number and percentage of patients with hemolytic events will be summarized by preferred term, severity (based on CTCAE grades), type of adverse event, relation to study treatment by the phases or subsets previously described.
Evaluate gastrointestinal events for study period. | 104 weeks
  The number and percentage of patients with gastrointestinal events will be summarized by preferred term, severity (based on CTCAE grades), type of adverse event, relation to study treatment by the phases or subsets previously described.
Evaluate the proportion of patients still in MR4 (BCR-ABL ≤ 0.01%) within 52 weeks following ponatinib therapy cessation. | 52 weeks
  Number of patients still in MR4 and have not restarted TKI therapy in the first 52 weeks after starting ponatinib TFR phase divided by the number of patients who entered ponatinib TFR phase.
Evaluate the proportion of patients still in MMR within 24 weeks following ponatinib therapy cessation. | 24 weeks
  The number of patients who still have a MMR and have not restarted TKI therapy in the first 24 weeks after starting ponatinib TFR phase divided by the number of patients who entered ponatinib TFR phase.
To estimate progression-free survival (PFS) | 4 years
  Time from start ponatinib treatment to the occurrence of progression to AP/BC, loss of MMR or death from any cause, the earliest of these events.
Treatment-free survival (TFS) | 104 weeks
  time from ponatinib cessation to the occurrence of loss of MMR, restart of TKI treatment, progression of AP/BC, or death from any cause, the earliest of these events.

OTHER OUTCOMES:
Evaluate the proportion of patients who achieve a MR 5 at ponatinib therapy cessation. | 104 weeks
  The number of patients who achieve a MR 5 at ponatinib therapy cessation divided by the number of patients who entered ponatinib TFR phase.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Martínez López, MD, Principal Investigator — Hospital Universitario 12 de Octubre; Valentín García Gutierrez, MD, Principal Investigator — Hospital Universitario Ramon y Cajal; Juan Carlos Hernández Boluda, MD, Principal Investigator — Hospital Clínico de Valencia
Locations (13):
- Spain (13):
  - Institut Català D'Oncologia L'Hospitalet (ICO), L'Hospitalet de Llobregat, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid, Madrid
  - Hospital Ramón y Cajal, Madrid, Madrid
  - Hospital Universitario y Politécnico La Fe, Valencia, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia, Valencia
  - Institut Català d´oncologia Badalona (ICO), Badalona
  - Hospital Universitario de Gran Canaria Dr. Negrín, Las Palmas de Gran Canaria
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Complejo Hospitalario Regional de Málaga, Málaga
  - Hospital Virgen de La Victoria, Málaga
  - Hospital General Universitario J.M. Morales Meseguer, Murcia
  - Hospital Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No